CLINICAL TRIAL: NCT05395702
Title: Pilot Single-center Open Study of the Effect of Ingaron on the Efficacy and Resistance to Antibiotics in Antibacterial Therapy in Patients With Community-acquired Pneumonia
Brief Title: Study of Ingaron's Effect on Efficacy and Resistance to Antibiotics in Community-acquired Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPP Pharmaclon Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN/100000-317
Record Dates: First submitted 2022-05-19; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Community-acquired Pneumonia
Keywords: interferon gamma; IFN-g; antibiotic resistance; Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Interferon-gamma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: Interferon Gamma (Experimental): Antibacterial therapy + IFN-G administered intramuscularly 100,000 IU once a day daily for 5 days
  Interventions: Drug: Interferon-Gamma
- Control: No intervention (No Intervention): Only antibacterial therapy

INTERVENTIONS:
Drug: Interferon-Gamma — received by microbiological synthesis; specific antiviral activity on cells is 2x10*7 Units per mg of protein
  Other Names: Ingaron; Interferon gamma human recombinant
  Arms: Drug: Interferon Gamma

SUMMARY:
The primary purpose of this study is to effect of Ingaron®, a lyophilisate for the preparation of a solution for intramuscular and subcutaneous administration of 100,000 IU (LLC NPP Farmaklon, Russia) on the effectiveness of antibiotic therapy in patients with community-acquired pneumonia who fell ill during the epidemiological rise of ARVI.

DETAILED DESCRIPTION:
Pilot, open, single-centre, randomized controlled trial. Patients will be prescribed basic combination antibiotic therapy. In addition to antibiotic therapy, half of the patients will receive Ingaron®, a lyophilisate for the preparation of a solution for intramuscular and subcutaneous administration of 100,000 IU (LLC NPP Farmaklon, Russia). The study drug solution Ingaron® will be administered intramuscularly at 100,000 IU once daily for 5 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of the inpatient department of both sexes aged 18 to 60 years.
2. Confirmed diagnosis - community-acquired pneumonia (causative agent not specified) of an uncomplicated typical course without respiratory failure and the duration of symptoms is not more than 14 days.
3. Risk class of lethal outcome I-II according to the Fine scale.
4. Availability of an Informed Consent voluntarily signed by the patient.

Exclusion Criteria:

1. Increased individual sensitivity to gamma interferon, Ingaron® and / or excipients that are part of Ingaron® or drugs used in antibacterial therapy.
2. The use of immunomodulating, immunostimulating or immunosuppressive therapy later than 1 month before enrollment in the study.
3. Bronchial asthma and/or COPD.
4. Congestive heart failure.
5. Acute diseases of the gastrointestinal tract or other pathologies that may affect the absorption, distribution, metabolism or excretion of drugs.
6. Chronic liver and / or kidney disease or other pathologies that may affect the absorption, distribution, metabolism or excretion of drugs.
7. Oncological diseases, autoimmune, immunosuppressive conditions at present or according to history.
8. Cerebrovascular pathologies.
9. Diabetes.
10. Pregnancy or lactation.
11. Smoking index over 10 pack/years.
12. Data on severe nervous or mental diseases, including history.
13. Violation of consciousness.
14. Participation of the patient in other studies with the use of drugs or other methods of therapy, including clinical, currently or later than 1 month before inclusion in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Time to clinical stabilization of the patient's condition | Day 33
  Assessed by the following parameters: HR < 100 bpm, RR < 24 resp./min, systolic blood pressure ≥90 mmHg, blood saturation level ≥ 90%

SECONDARY OUTCOMES:
Change in the level of procalcitonin in the blood | Day 10
  Change in the level of procalcitonin in the blood at visit 4 relative to visit 0
Change in the level of C-reactive protein in the blood | Day 10
  Change in the level of C-reactive protein in the blood at visit 4 relative to visit 0
Change in blood oxygen saturation | Day 3
  Change in blood oxygen saturation at visit 2 relative to visit 0
Change in blood oxygen saturation | Day 6
  Change in blood oxygen saturation at visit 3 relative to visit 0
Change in blood oxygen saturation | Day 10
  Change in blood oxygen saturation at visit 4 relative to visit 0
Borg Scale changes | Day 10
  Changes on the Borg Scale at visit 4 relative to visit 0, where the minimum score is 0 - dyspnea does not bother, the maximum score is 10 - dyspnea is very pronounced
Borg Scale changes | Day 31
  Changes on the Borg Scale during a phone call relative to visit 0, where the minimum score is 0 - shortness of breath does not bother, the maximum score is 10 - shortness of breath is very pronounced
Change in the volume of infiltrates in the lungs according to X-ray data | Day 10
  Change in the volume of infiltrates in the lungs according to X-ray data at visit 4 relative to visit 0
Difference between body temperature values | Day 3
  Difference between body temperature values
  Difference between body temperature values (in case of symptom presence according to screening data) at visit 2 relative to visit 0
Difference between body temperature values | Day 6
  Difference between body temperature values (in case of symptom presence according to screening data) at visit 3 relative to visit 0
Difference between body temperature values | Day 10
  Difference between body temperature values (in case of symptom presence according to screening data) at visit 4 relative to visit 0
Change in the level of leukocytes in the blood | Day 3
  Change in the level of leukocytes in the blood at visit 2 relative to visit 0
Change in the level of leukocytes in the blood | Day 10
  Change in the level of leukocytes in the blood at visit 4 relative to visit 0
ESR change | Day 10
  ESR change at visit 4 relative to visit 0
Change in bacterial count in sputum culture | Day 10
  Change in bacterial count in sputum culture at visit 4 relative to visit 0
Proportion of patients with antibiotic therapy failure | Day 3
  Proportion of patients with antibiotic therapy failure, assessed by the need to change the therapy regimen (add drugs, replace them, or switch to a different dosing regimen or route of administration), lack of signs of clinical stabilization of the condition, or worsening of the course of pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly I Saulin, Master, Study Director — SPP Pharmaclon Ltd.
Locations (1):
- City Clinical Hospital named after M.E. Zhadkevich Moscow City Health Department, Moscow, Russia

REFERENCES:
- [Result] Belevsky AS, Berns SA, Lartseva OA, Myasnikov AL, Nadaraya VM, Talyzin PA. Efficacy and safety of interferon gamma in the treatment of community-acquired pneumonia: results of an open-label randomized trial IN/100000-317. Meditsina. 2019; 4: 110-25.